CLINICAL TRIAL: NCT01910935
Title: Effectiveness of Physical Activity Prescription Among Hypertensive Patients of Primary Health Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-785-038; FIS/IMSS/PROT/G10/841 (Other: FIS/IMSS)
Record Dates: First submitted 2013-07-05; First posted 2013-07-30 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
Keywords: Physical activity; Hypertension; Scheme reference; Primary care
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity prescription (Experimental): 24 weeks physical activity program. 1 hour, 3 times a week, moderate to vigorous intensity.
  Interventions: Behavioral: Physical activity prescription to develop program in group.
- No physical activity prescription (No Intervention): Provide information to patients about the benefits of physical activity and how to increase it safely.

INTERVENTIONS:
Behavioral: Physical activity prescription to develop program in group. — Overall the intervention involves a medical reference in primary care (PHC) to hypertensive patients (during routine consultation) to assist the sports facilities of the same Institute, to develop a group program of physical activity which will last 24 weeks. Led by the trained staff in physical activity to patients with chronic diseases.
  Arms: Physical activity prescription

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a program to increase the physical activity of hypertensive patients using medical services and sports facilities of the Mexican Social Security Institute. The primary hypothesis to be proven is: The intervention will increase the proportion of hypertensive patients complying the physical activity minimum at week to get benefits on health in 20%, compare to patients in control group.

DETAILED DESCRIPTION:
Secondary Hypothesis:

The intervention achieved a significant change in the group of hypertensive patients in the following variables:

1. Decreased levels of systolic and diastolic blood pressure, biochemical markers such as total cholesterol, triglycerides and fasting blood glucose and increased HDL cholesterol.
2. Increase muscular endurance and cardio-respiratory capacity according to the categories of risk stratification.
3. Decreased body weight, body mass index and waist circumference.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with high blood pressure <5 years of evolution and / or without use of drug therapy to treat that condition;
* with low levels of physical activity (PA) or physically inactive (less than 150 minutes of PA at week, intensity moderate to vigorous);
* with availability to PA practice or considering begin to PA practice within the next six months (contemplation or preparation stages of the Transtheoretical Model).
* Without cardiovascular risk (assessed previously);
* Without physical or mobility problems that impede PA practice;
* Willingness to participate in the study, fulfill with outlined activities to develop the proposal.

Exclusion Criteria:

* high-risk patients according to the risk stratification of the American College of Sports Medicine;
* fulfill the high recommendation of physical activity (more than 300 minutes per week of moderate to vigorous intensity);

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Physical activity. Level of physical activity between intervention and control groups. | 24 weeks
  The length of the intervention is 24 weeks, the control group will be followed for 24 weeks also. The outcome measure is a composite at three moments of the study. Basal measurement, 24 weeks and 36 weeks, this last moment to assess sustainability of the intervention.
  The intervention will be effective if the difference in the percent of population (complying the minimum recommended of physical activity) among control and intervention groups is at least of 20%.

SECONDARY OUTCOMES:
Blood pressure | 24 weeks
  Blood pressure among intervention and control groups, at the three moments of the study: basal measurement, 24 weeks (end of the intervention) and 36 weeks. The outcome measure is a composite at three moments of the study. Basal measurement, 24 weeks and 36 weeks, this last moment to assess sustainability of the intervention.

OTHER OUTCOMES:
Composite measure of biochemical markers: total cholesterol, triglycerides and fasting blood glucose | 24 weeks
  Biochemical markers (total cholesterol, triglycerides and fasting blood glucose) among intervention and control groups, at the three moments of the study: basal measurement, 24 weeks (end of the intervention) and 36 weeks. The secondary outcome measure is a composite at three moments of the study. Basal measurement, 24 weeks and 36 weeks, this last moment to assess sustainability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gallegos-Carrillo Katia, D. Sc, Principal Investigator — Instituto Mexicano del Seguro Social/Unidad de Investigación Epidemiologica y en Servicios de Salud.
Locations (1):
- Instituto Mexicano del Seguro Social. Morelos. HGR/MF. No, UMF 3, UMF 20, UMF 23, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Derived] Gallegos-Carrillo K, Garcia-Pena C, Salmeron J, Salgado-de-Snyder VN, Vazquez-Cabrer G, Lobelo F. Exercise-referral scheme to promote physical activity among hypertensive patients: design of a cluster randomized trial in the Primary Health Care Units of Mexico's Social Security System. BMC Public Health. 2014 Jul 9;14:706. doi: 10.1186/1471-2458-14-706. PMID 25011612